CLINICAL TRIAL: NCT06404996
Title: Smart-phone Application Versus Conventional Paper for the Documentation of Voiding Dysfunction in Children: Which Diary is Most Advantageous
Brief Title: Smart-phone Application Versus Conventional Paper for the Documentation of Voiding Dysfunction in Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah International Medical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB/0550/24
Record Dates: First submitted 2024-04-22; First posted 2024-05-08 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Voiding Dysfunction; Children
Keywords: voiding dysfunction; bladder; children; voiding diary; smart-phone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smart-phone diary (Experimental): smart-phone voiding diary application
  Interventions: Device: Smart-phone Voiding Diary
- Paper diary (Active Comparator): Conventional paper based voiding diary
  Interventions: Diagnostic Test: Paper voiding diary

INTERVENTIONS:
Device: Smart-phone Voiding Diary — Smart-phone Voiding Diary
  Other Names: DryDawn
  Arms: Smart-phone diary
Diagnostic Test: Paper voiding diary — Conventional Paper voiding diary
  Arms: Paper diary

SUMMARY:
The objective of the research is to compare the written voiding diary method to the smart-phone diary, DryDawn®, which the investigators selected among several applications using specific criteria appropriate to our population. The investigators aim is to describe the method that proves to be most efficient by assessing which diary provides the best quality and amount of information, and draws the highest level of satisfaction from participants.

Patient satisfaction will be assessed using a questionnaire that was designed for use in this study.

DETAILED DESCRIPTION:
The idea of using smart-phone applications for the purpose of medical management is not new, however, results from studies have been variable and few have characterized their use in the management of disease in children. The propose of study is to conduct a a research that involves the use of a smart-phone voiding diary application in children.

The intention of this research is to identify which method of documentation, either a smart-phone voiding diary application or the conventional written diary, is most effective in gathering information from urology patients in the pediatric population.

The investigators will conduct a prospective randomized study to investigate which type of diary is better regarding data collection and patient's satisfaction. Consenting individuals will be informed of the study details and their safety will be assured. Patients/parents will be informed of their right to withdraw from the study at any moment.

The two groups refer to the two methods of documentation (diaries) to which will be randomly assigned .The diaries are the smart-phone diary application, DryDawn ® (The Arabic version), or the conventional pen-and-paper method.

A website (www.randomizer.org) will be used to generate a randomized numbered lists that determine participant allocation to one of two study groups.

Data collection will include patient demographics, the type of diary used, as well as the information that participants provide in either of the voiding the diaries and the satisfaction questionnaire. The investigators will analyze the data and report on the percentage of participants who complied with their diary completion, information provided by patients and caregivers in the diary, and the number of participants in the study. Moreover, a questionnaire (Voiding diary Satisfaction Questionnaire) will be given to each family evaluating the patient/caregiver satisfaction.

If the diary has to be repeated, automatically will switch to the other type of diary. A re-evaluation of the diary satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* New patients who have a voiding dysfunction that necessitates the use of a voiding diary
* Children ages six (6) to eighteen (18) years
* Participants must own a smart-phone

Exclusion Criteria:

* Children less than six (6) years of age
* Participants who do not own a smart-phone

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
The percentage of diary completion | 1 year
  The percentage/number of patients of each group who will complete the diary and send it on-time.

SECONDARY OUTCOMES:
Patient's satisfaction assessment by the Voiding diary Satisfaction Questionnaire | 1 year
  Patient satisfaction will be assessed using a Voiding diary Satisfaction Questionnaire that can assess the ease of use of the diary chosen, as well as the compliance of diary completion and submission. The questionnaire consists of 6 subjective questions. Each question has 2-5 different answers with no objective scale.

CONTACTS AND LOCATIONS:
Overall Officials: Amr Hodhod, MD, PhD, Msc, Principal Investigator — King Abdullah International Medical Research Center

IPD SHARING:
Plan to Share IPD: No
Because of data ownership policy of our institution, I may not able to share full data unless approved by the ethical committee